CLINICAL TRIAL: NCT00376597
Title: A Randomized Study to Prevent Lymphedema in Women Treated for Breast Cancer
Brief Title: Education With or Without Exercise and Counseling in Preventing Lymphedema in Women With Stage I, Stage II, or Stage III Breast Cancer Who Are Undergoing Axillary Lymph Node Dissection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CALGB-70305; CDR0000494652 (Registry Identifier: NCI Physician Data Query); NCI-2009-00488 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA037447 (NIH)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-01

CONDITIONS: Lymphedema
Keywords: lymphedema; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Early Intervention, Educational; Methods; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lymphedema education) (Experimental): Six weeks after surgery, patients receive a brief initial post-operative care session describing lymphedema risk and prevention through oral instruction and written materials. Patients complete physical assessments and questionnaires at 6 weeks and at 6, 12, and 18 months. Patients are also contacted by telephone at 9 and 15 months.
  Interventions: Other: quality of life assessment; Other: educational intervention
- Arm II (lymphedema education, physical therapy) (Experimental): Description Patients receive lymphedema education and complete physical assessments and questionnaires as in Arm I. Patients also complete a personalized physical therapy intervention, receive a refrigerator magnet, and a 15-minute video that reinforces information and exercises.
  Interventions: Other: quality of life assessment; Other: educational intervention; Procedure: Physical therapy

INTERVENTIONS:
Other: quality of life assessment — Ancillary studies
Other: educational intervention — Receive lymphedema educational materials
  Other Names: intervention, educational
Procedure: Physical therapy — Complete physical therapy-focused intervention
  Other Names: physiotherapy
  Arms: Arm II (lymphedema education, physical therapy)

SUMMARY:
This randomized phase III trial studies how well education with or without physical therapy intervention works in preventing lymphedema in women with stage I, II, or III breast cancer who are undergoing axillary lymph node dissection (surgery to remove lymph nodes found in the armpit region). Lymphedema is a condition in which extra lymph fluid builds up in tissues and causes swelling in an arm or leg if lymph vessels are blocked, damaged, or removed by surgery. A personalized physical therapy intervention and education materials may be better than education materials alone in preventing lymphedema in women with breast cancer who are undergoing axillary lymph node dissection.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To test, in a group randomized controlled trial, the efficacy of this program versus education only in reducing the incidence of lymphedema.

II. To compare the severity of lymphedema, in terms of changes in arm circumference at the site of greatest difference as a continuous variable between the two interventions.

III. To assess the agreement between patients' self-report of swelling (mild, moderate, and severe) and the extent of circumferential measurement difference between the treated side and the contralateral arm at the site of greatest difference.

IV. To compare the health-related quality of life (Factional Assessment of Cancer Therapy-Breast [FACT-B]+4 score) between the two interventions.

V. To characterize adherence to lymphedema prevention exercises, lymphedema knowledge, and range of motion.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Six weeks after surgery, patients receive a brief initial post-operative care session describing lymphedema risk and prevention through oral instruction and written materials. Patients complete physical assessments and questionnaires at 6 weeks and at 6, 12, and 18 months. Patients are also contacted by telephone at 9 and 15 months.

ARM II: Patients receive lymphedema education and complete physical assessments and questionnaires as in Arm I. Patients also complete a personalized physical therapy intervention, receive a refrigerator magnet, and a 15-minute video that reinforces information and exercises.

ELIGIBILITY:
Eligibility Criteria:

* Newly diagnosed with stage I-III cancer of the female breast
* No prior history of carcinoma in situ, lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS), or invasive breast cancer

  * Patients with a history of other invasive malignancies are eligible as long as they have completed treatment and are 5 years post-diagnosis; patients with basal cell and squamous cell cancer of the skin are eligible
* Neoadjuvant therapy

  * Patients scheduled to receive any type of radiation therapy to the breast or axilla are eligible; however, they must be registered to this study with pre-surgery measures taken prior to receiving neoadjuvant therapy
  * Patients scheduled to receive neoadjuvant chemotherapy are also eligible; however, they must be registered to this study with pre-surgery measurements taken prior to receiving neoadjuvant therapy
  * Patients receiving no neoadjuvant therapy are eligible
* May be enrolled on other treatment trials; however, patients enrolled on surgery trials where only one treatment arm is full axillary node dissection are not eligible; NOTE: Patients enrolled on American College of Surgeons Oncology Group (ACOSOG)-Z1071 are eligible to participate in this study; patients concurrently enrolled on this study and ACOSOG-Z1071, may not also be enrolled on the ACOSOG-Z1071 lymphedema sub-study
* No documented cardiac conduction disturbances, unstable angina, dementia, or any other chronic disease which, in the opinion of the treating physician, significantly increases mortality over the next 2 years
* No diagnosed lymphedema
* In order to be properly fitted for the elastic sleeve, eligible patients must have arm measurements for axilla, elbow, and wrist that fall within the ranges for one of the six sleeve sizes
* Not currently homebound or dependent upon a walker or wheelchair for mobility
* Able to participate in a mild exercise program
* Willing to return to the study site for the duration of the study (18 months)
* Sentinel (SND) or full axillary node dissection (AND) (no minimum number of nodes required)
* Patients with double mastectomy, axillary node dissection and/or radiation on both arms are ineligible; patients who undergo these treatments (i.e., surgery and/or radiation) on the contralateral arm after registration to Step 2 are still eligible to remain in the study; however, it should be documented appropriately on form C-1628 at the conclusion of study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Electra D. Paskett, PhD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (76):
- United States (76):
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Valley Medical Oncology, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Kaiser Permanente at Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - North Broward Medical Center, Deerfield Beach, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Bettendorf, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Kaiser Permanente at Woodlawn Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Kaiser Permanente - Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center Cancer Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Trinitas Comprehensive Cancer Center at Trinitas Hospital, Elizabeth, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Kaiser Permanente Medical Center - Fair Oaks, Fairfax, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia

REFERENCES:
- [Derived] Paskett ED, Le-Rademacher J, Oliveri JM, Liu H, Seisler DK, Sloan JA, Armer JM, Naughton MJ, Hock K, Schwartz M, Unzeitig G, Melnik M, Yee LD, Fleming GF, Taylor JR, Loprinzi C. A randomized study to prevent lymphedema in women treated for breast cancer: CALGB 70305 (Alliance). Cancer. 2021 Jan 15;127(2):291-299. doi: 10.1002/cncr.33183. Epub 2020 Oct 20. PMID 33079411
- [Derived] Naughton MJ, Liu H, Seisler DK, Le-Rademacher J, Armer JM, Oliveri JM, Sloan JA, Hock K, Schwartz M, Unzeitig G, Melnik M, Yee LD, Fleming GF, Taylor JR, Loprinzi C, Paskett ED. Health-related quality of life outcomes for the LEAP study-CALGB 70305 (Alliance): A lymphedema prevention intervention trial for newly diagnosed breast cancer patients. Cancer. 2021 Jan 15;127(2):300-309. doi: 10.1002/cncr.33184. Epub 2020 Oct 20. PMID 33079393

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Lymphedema Education, Physical Therapy): Patients receive lymphedema education and complete physical assessments and questionnaires as in Arm I. Patients also complete a personalized physical therapy intervention, receive a refrigerator magnet, and a 15-minute video that reinforces information and exercises.
Period: Overall Study
Arm/Group | Arm I (Lymphedema Education) | Arm II (Lymphedema Education, Physical Therapy)
Started | 253 | 315
Completed | 242 | 312
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Population: 554 patients were treated and analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lymphedema Education) | Arm II (Lymphedema Education, Physical Therapy) | Total
Number analyzed (Participants) | 242 | 312 | 554
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.4) | 57.5 (11.2) | 57.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 312 | 554
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 242 | 312 | 554

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Lymphedema-free 18 Months After Randomization
Description: To test, in a group randomized controlled trial, the efficacy of this program versus education only in reducing the incidence of lymphedema. Reported here is the proportion of patients who are lymphedema-free 18 months after randomization between the two arms
Time Frame: 18 months
Population: 554 patients completed treatment and were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lymphedema Education) | Arm II (Lymphedema Education, Physical Therapy)
Number analyzed (Participants) | 242 | 312
Participants | 114 | 135

2. Secondary Outcome: Change From Baseline at 18 Months in Arm Circumference at the Site of Greatest Difference
Description: To compare the severity of lymphedema in terms of changes in arm circumference at the site of greatest difference as a continuous variable between the two interventions.
Time Frame: 18 months
Population: 402 patients were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: cubic cm
Arm/Group | Arm I (Lymphedema Education) | Arm II (Lymphedema Education, Physical Therapy)
Number analyzed (Participants) | 182 | 220
cubic cm | 55.1 (333.3) | 46.6 (417.2)

3. Secondary Outcome: Agreement Between Patients' Self-report of Swelling and the Extent of Circumferential Measurement Difference Between the Treated Side and the Contralateral Arm
Description: To assess the agreement between patients' self-report of swelling (mild, moderation and severe) and the extent of circumferential measurement difference between treated side and the contralateral arm at the site of greatest difference. Per protocol, this analysis will include all patients and not be comparing the intervention arm with the control arm.
Time Frame: 18 months
Population: 368 patients filled out a self assessment of swelling and were analyzed. This includes all patients that filled out a self-report of swelling, the two arms are combined because this is a comparison of actual swelling against self reported swelling, not a comparison of interventions.
Measure: Count of Participants; unit: Participants
Groups:
- All Treated Patients: This Arm consists of both Arm I and Arm II.
Arm/Group | All Treated Patients
Number analyzed (Participants) | 368
Participants
  <0.5in difference between arms: number analyzed (Participants) | 363
  <0.5in difference between arms: Self Report None/Mild Swelling | 353
  <0.5in difference between arms: Self Report Moderate swelling | 8
  <0.5in difference between arms: Selft Report Severe swelling | 2
  0.5in - 2in difference between arms: number analyzed (Participants) | 11
  0.5in - 2in difference between arms: Self Report None/Mild Swelling | 11
  0.5in - 2in difference between arms: Self Report Moderate swelling | 0
  0.5in - 2in difference between arms: Selft Report Severe swelling | 0
  >= 2in difference between arms: number analyzed (Participants) | 2
  >= 2in difference between arms: Self Report None/Mild Swelling | 1
  >= 2in difference between arms: Self Report Moderate swelling | 1
  >= 2in difference between arms: Selft Report Severe swelling | 0

4. Secondary Outcome: Health-related Quality of Life as Assessed by FACT-B +4 Score
Description: To compare the health-related quality of life (FACT-B+4 score) between the two interventions. The change between baseline and month 18 for the total plus 4 score will be reported here. The total plus 4 score is an average of the physical, social, emotional, functional, FACT-G, and additional concerns sub-scales. Each sub-scale has questions ranging from 1-5. Once the average of all subscales is taken, the total plus 4 score is converted into a score out of 100. 100 being the best, 0 being the worst.
Time Frame: 18 months
Population: 326 patients were analyzed for this measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm I (Lymphedema Education) | Arm II (Lymphedema Education, Physical Therapy)
Number analyzed (Participants) | 142 | 184
Units on a scale | 1.4 (8.6) | 0.1 (8.9)

5. Secondary Outcome: Adherence to Lymphedema Prevention Exercises, Lymphedema Knowledge, Range of Motion, and Arm Strength
Description: To characterize adherence to lymphedema prevention exercises, lymphedema knowledge and range of motion. The frequency of elastic sleeve use for heavy arm use/exercise/air travel will be reported here. Arm I did not receive a sleeve to wear, thus will not be reported.
Time Frame: from baseline up to 18 months
Population: 236 patients were analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (Lymphedema Education, Physical Therapy)
Number analyzed (Participants) | 236
Participants
  6 months: >=75% | 77
  6 months: 1%-74% | 108
  6 months: Not at all/never | 51
  12 months: number analyzed (Participants) | 209
  12 months: >=75% | 66
  12 months: 1%-74% | 94
  12 months: Not at all/never | 49
  18 months: number analyzed (Participants) | 214
  18 months: >=75% | 67
  18 months: 1%-74% | 92
  18 months: Not at all/never | 55

ADVERSE EVENTS:
Time Frame: No adverse events were collected
Arm/Group | Arm I (Lymphedema Education) | Arm II (Lymphedema Education, Physical Therapy)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less